CLINICAL TRIAL: NCT06739421
Title: The Diagnostic Value of Bronchoscopic Needle-based Confocal Laser Endomicroscopy (nCLE) As a Real-time Detection Tool for Diagnosing Peripheral Lung Cancer: a Multi-centre Randomised Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Professor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022YFC2404404-PN
Record Dates: First submitted 2024-12-17; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer, Non-Small Cell; Lung Cancer, Small Cell
Keywords: needle-based confocal laser endomicroscopy; peripheral lung cancer; peripheral lung nodules; lung biopsy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- nCLE-NB-rEBUS-forcep biopsy (Experimental): The participants would undergo lung biopsy using forcep, under the guidance of bronchoscopic needle-based confocal laser endomicroscopy (nCLE) with the assistance of navigation bronchoscopy (NB) and radial endobronchial ultrasound (rEBUS)
  Interventions: Procedure: nCLE-NB-rEBUS-forcep biopsy
- nCLE-NB-rEBUS-TBCB (Experimental): The participants would undergo transbronchial crybiopsy (TBCB) , under the guidance of bronchoscopic needle-based confocal laser endomicroscopy (nCLE) with the assistance of navigation bronchoscopy (NB) and radial endobronchial ultrasound (rEBUS)
  Interventions: Procedure: nCLE-NB-rEBUS-TBCB
- NB-rEBUS-forcep biopsy (Active Comparator): The participants would undergo lung biopsy using forcep, under the guidance of navigation bronchoscopy (NB) and radial endobronchial ultrasound (rEBUS)
  Interventions: Procedure: NB-rEBUS-forcep biopsy
- NB-rEBUS-TBCB (Active Comparator): The participants would undergo transbronchial crybiopsy (TBCB) , under the guidance of navigation bronchoscopy (NB) and radial endobronchial ultrasound (rEBUS)
  Interventions: Procedure: NB-rEBUS-TBCB

INTERVENTIONS:
Procedure: nCLE-NB-rEBUS-forcep biopsy — The participants would undergo lung biopsy using forcep, under the guidance of bronchoscopic needle-based confocal laser endomicroscopy (nCLE) with the assistance of navigation bronchoscopy (NB) and radial endobronchial ultrasound (rEBUS)
  Arms: nCLE-NB-rEBUS-forcep biopsy
Procedure: nCLE-NB-rEBUS-TBCB — The participants would undergo transbronchial crybiopsy (TBCB), under the guidance of bronchoscopic needle-based confocal laser endomicroscopy (nCLE) with the assistance of navigation bronchoscopy (NB) and radial endobronchial ultrasound (rEBUS)
  Arms: nCLE-NB-rEBUS-TBCB
Procedure: NB-rEBUS-forcep biopsy — The participants would undergo lung biopsy using forcep, under the guidance of navigation bronchoscopy (NB) and radial endobronchial ultrasound (rEBUS)
  Arms: NB-rEBUS-forcep biopsy
Procedure: NB-rEBUS-TBCB — The participants would undergo transbronchial crybiopsy (TBCB), under the guidance of navigation bronchoscopy (NB) and radial endobronchial ultrasound (rEBUS)
  Arms: NB-rEBUS-TBCB

SUMMARY:
The goal of this prospective, multi-centre, randomised controlled clinical study is to evaluate the diagnostic efficacy and safety of nCLE guided lung biopsy in patients with for peripheral lung nodules under the assistance of navigation bronchoscopy (NB) and radial endobronchial ultrasound (rEBUS), and assess whether the biopsy techniques, namely transbronchial crybiopsy (TBCB) and transbronchial forceps biopsy (TBFB), would influence the diagnostic efficacy and safety of nCLE guided biopsy.

Participants will divided into nCLE-NB-rEBUS-forcep biopsy group, nCLE-NB-rEBUS-TBCB group, NB-rEBUS-forcep biopsy group, and NB-rEBUS-TBCB group at a 1:1:1:1 ratio by using central, computerized random sequence, and then undertake nCLE-NB-rEBUS-forcep biopsy, nCLE-NB-rEBUS-TBCB, NB-rEBUS-forcep biopsy, and NB-rEBUS-TBCB according to the group.

Researchers will compare the diagnostic yield and incidence of adverse events of the four biopsy techniques.

ELIGIBILITY:
Inclusion Criteria:

* patients with peripheral lung nodules suspected of lung cancer based on CT scan (10mm≤size<30mm);
* patients requiring diagnostic bronchoscopy procedure to determine the benign or malignant nature of the lung nodule;
* Patients who can understand the purpose of the trial, participate voluntarily and sign an informed consent form.

Exclusion Criteria:

* Inability or non-willingness to provide informed consent;
* Endobronchial visible malignancy on bronchoscopic inspection;
* Target lesion within reach of the linear EBUS scope;
* Failure to comply with the study protocol;
* Known allergy or risk factors for an allergic reaction to fluorescein;
* Pregnancy or breast feeding;
* Haemodynamic instability;
* Refractory hypoxaemia;
* Therapeutic anticoagulant use that cannot be withheld for an appropriate interval before the procedure;
* Unable to tolerate general anaesthesia according to the anaesthesiologist;
* Undergoing chemotherapy as several chemotherapies have fluorescent properties at the same wavelength (eg, doxorubicin).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic yield of lung forcep biopsy and TBCB under guidance of nCLE-NB-rEBUS | 7 days after the biopsy
  The proportion of participants in whom the biopsy led to a definitive diagnosis.
Sensitivity of lung forcep biopsy and TBCB under guidance of nCLE-NB-rEBUS | 7 days after the biopsy
  The proportion of participants of lung cancer in whom the biopsy led to a definitive diagnosis .

SECONDARY OUTCOMES:
Incidence rate of adverse events | 7 days after the biopsy
  Symptoms and signs
the adequacy of sample acquisition | 7 days after the biopsy
  Samples resulting in a specific diagnosis or samples with the presence of lymphpcytes were considered as adequate.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, , 100029, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided